CLINICAL TRIAL: NCT00454818
Title: A Phase 1/2 Trial of Intracoronary Administration of MYDICAR® (AAV1/SERCA2a) in Subjects With Heart Failure in Two Stages (Open-Label, Sequential Dose-Escalation Cohorts and Randomized, Double-Blind, Placebo-Controlled, Parallel Cohorts)
Brief Title: Efficacy and Safety Study of Genetically Targeted Enzyme Replacement Therapy for Advanced Heart Failure
Acronym: CUPID
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celladon Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELL-001; CUPID Trial (Registry Identifier: NCT00454818)
Record Dates: First submitted 2007-03-30; First posted 2007-04-02 (Estimated); Results first posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Heart Failure, Congestive; Dilated Cardiomyopathy
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- MYDICAR Very Low Dose (Experimental): Single dose of MYDICAR, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1.4x10e11 DNAase resistant particles administered by antegrade epicardial coronary artery infusion. Used in MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study) only.
  Interventions: Genetic: MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study)
- MYDICAR Low Dose (Experimental): Single dose of MYDICAR, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 6x10e11 DNAase resistant particles administered by antegrade epicardial coronary artery infusion. Used in MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study) and MYDICAR Phase 2 (Placebo-controlled, Randomized Study)
  Interventions: Genetic: MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study); Genetic: MYDICAR Phase 2 (Placebo-controlled, Randomized Study)
- MYDICAR Mid Dose (Experimental): Single dose of MYDICAR, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 3x10e12 DNAase resistant particles administered by antegrade epicardial coronary artery infusion. Used in MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study) and MYDICAR Phase 2 (Placebo-controlled, Randomized Study).
  Interventions: Genetic: MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study); Genetic: MYDICAR Phase 2 (Placebo-controlled, Randomized Study)
- MYDICAR High Dose (Experimental): Single dose of MYDICAR, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1x10e13 DNAase resistant particles administered by antegrade epicardial coronary artery infusion. Used in MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study) and MYDICAR Phase 2 (Placebo-controlled, Randomized Study).
  Interventions: Genetic: MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study); Genetic: MYDICAR Phase 2 (Placebo-controlled, Randomized Study)
- Placebo infusion (Placebo Comparator): A single dose of placebo (Sodium Chloride Injection, USP) administered by antegrade epicardial coronary artery infusion.
  Interventions: Procedure: Placebo Infusion

INTERVENTIONS:
Genetic: MYDICAR Phase 1 (Open-label, Serial Dose-Escalation Study) — MYDICAR administered by antegrade epicardial coronary artery infusion
  Other Names: AAV1/SERCA2a
  Arms: MYDICAR High Dose; MYDICAR Low Dose; MYDICAR Mid Dose; MYDICAR Very Low Dose
Procedure: Placebo Infusion — Saline; epicardial coronary artery infusion
  Arms: Placebo infusion
Genetic: MYDICAR Phase 2 (Placebo-controlled, Randomized Study) — MYDICAR administered by antegrade epicardial coronary artery infusion
  Other Names: AAV1/SERCA2a
  Arms: MYDICAR High Dose; MYDICAR Low Dose; MYDICAR Mid Dose

SUMMARY:
The study is divided into 2 parts. In the first part, the safety of the gene transfer agent MYDICAR® will be evaluated. In the second part, the ability of MYDICAR® to improve heart function will be studied.

DETAILED DESCRIPTION:
The American Heart Association (AHA) 2006 update on heart disease reported that 5 million Americans are believed to have symptomatic heart failure (HF), and 550,000 patients are newly diagnosed each year. The estimated direct and indirect cost of HF in the United States (U.S.) for 2006 will be ~$29.6 billion. Heart failure is a disabling chronic disease and the most frequent discharge diagnosis for hospitalization among older adults. Despite the significant resources expended on the treatment of this disease, outcomes remain poor. The five-year survival for individuals diagnosed with heart failure is less than 50%, and in end-stage heart failure, the one-year survival may be as low as 25% regardless of medical therapy.

Recent studies suggest that the failing heart is not refractory to treatment, as was previously believed. For example, the observation that a small percentage of subjects with left ventricular assist devices (LVADs) can be permanently weaned from their device strongly suggests that damaged hearts are capable of recovering lost function.

Clinical studies of MYDICAR® have not yet been conducted in humans. Celladon Corporation (Celladon) proposes to investigate gene transfer as a method to restore SERCA2a function in heart failure (HF) patients using a recombinant adeno-associated viral vector (AAV), which consists of an AAV serotype 1 capsid and contains the human SERCA2a complementary DNA (cDNA) flanked by Inverted Terminal Repeats (ITR) derived from AAV serotype 2 (AAV1/SERCA2a). MYDICAR® refers to AAV1/SERCA2a drug product intended for administration by percutaneous delivery.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ischemic or non-ischemic cardiomyopathy. Subjects with ischemic cardiomyopathy must have at least one major coronary vessel with Thrombolysis in Myocardial Infarction (TIMI) grade 3 flow.
* Left ventricular ejection fraction (LVEF) ≤35%
* Diagnosis of New York Heart Association (NYHA) Class III/IV heart failure for a minimum of 3 months prior to screening
* Maximal oxygen consumption (VO2 max) ≤20 mL/kg/min within 90 days prior to enrollment
* An implantable cardioverter defibrillator (ICD) implanted a minimum of 30 days prior to enrollment
* Treatment with appropriate heart failure therapy as tolerated
* All women of childbearing potential must have a negative urine pregnancy test prior to administration of investigational product and agree to use adequate contraception. Men capable of fathering a child must agree to use barrier contraception or limit activity to post-menopausal, surgically sterilized, or a contraception-practicing partner, for 3 months after administration of investigational product.
* Ability to sign Informed Consent Form (ICF) and Release of Medical Information Form

Exclusion Criteria:

* Any intravenous therapy with positive inotropes, vasodilators, or diuretics within 30 days prior to enrollment
* Restrictive cardiomyopathy, obstructive cardiomyopathy, pericardial disease, amyloidosis, infiltrative cardiomyopathy, uncorrected thyroid disease, or dyskinetic LV aneurysm
* Cardiac surgery, percutaneous coronary intervention, or valvuloplasty within 30 days prior to enrollment
* Clinically significant myocardial infarction (e.g., ST elevation MI [STEMI] or large non-STEMI) within 6 months prior to enrollment
* Prior heart transplantation, left ventricular reduction surgery (LVRS), cardiomyoplasty, passive restraint device (e.g., CorCap™ Cardiac Support Device), surgically implanted LVAD or cardiac shunt
* Likely to receive cardiac resynchronization therapy, cardiomyoplasty, LVRS, heart transplant, conventional revascularization procedure, or valvular repair within 6 months following enrollment
* Patients with prior coronary artery bypass graft(s) (CABG) will reviewed on a case-by-case basis
* No evidence of functional or viable myocardium
* Exercise capacity primarily limited by obesity, peripheral vascular disease, intrinsic pulmonary disease or orthopedic problems and not by underlying heart failure
* Known hypersensitivity to octafluoropropane (component of the intravenous echocardiography contrast agent, DEFINITY®) or other contrast dyes used for angiography; history of, or likely need for, high dose steroid pretreatment prior to contrast angiography
* A left ventricle that is difficult to image or high quality echocardiography is not obtainable at screening
* Significant left main or ostial right coronary lumenal stenosis in the opinion of the investigator
* Expected survival <1 year in the investigator's medical opinion
* Suspected or active viral, bacterial, fungal, or parasitic infection within 48 hours prior to enrollment
* Liver function tests (alanine aminotransferase [ALT], aspartate aminotransferase [AST], alkaline phosphatase) >2x Upper Limit of Normal (ULN) within 30 days prior to enrollment or known intrinsic liver disease (e.g., cirrhosis, chronic hepatitis B or hepatitis C virus infection)
* Current or likely need for hemodialysis within 12 months following enrollment
* Bleeding diathesis or thrombocytopenia defined as platelet count <50,000 platelets/μL
* Anemia defined as hemoglobin <10 g/dL
* Known AIDS or HIV-positive status, or a previous diagnosis of immunodeficiency with an absolute neutrophil count <1000 cells/mm3
* Previous participation in a study of gene transfer
* Presence of neutralizing anti-AAV1 antibodies at titer ≥1:2 within 3 months of screening
* Receiving investigational intervention or participating in another clinical study within 30 days or within 5 half-lives of the investigational drug administration prior to enrollment
* Pregnancy or lactation
* Recent history of psychiatric disease (including drug or alcohol abuse) that is likely to impair subject's ability to comply with protocol-mandated procedures, in the opinion of the investigator
* Other concurrent medical condition(s) that, while not explicitly excluded by the protocol, could jeopardize the safety of the patient or objectives of the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2007-03; Primary Completion 2010-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Jaski, MD, Principal Investigator — San Diego Cardiac Center; Donna Mancini, MD, Principal Investigator — Columbia University Hospital; Randall Starling, MD, Principal Investigator — The Cleveland Clinic; Mariell Jessup, MD, Study Chair — University of Pennsylvania; Thomas Cappola, MD, ScM, Principal Investigator — University of Pennsylvania; Daniel Pauly, MD, Principal Investigator — Shands Hospital, University of Florida at Gainesville; Barry London, MD, Principal Investigator — University of Pittsburgh Medical Center; Barry Greenberg, MD, Principal Investigator — University of California at San Diego Medical Center; A. G. Kfoury, MD, Principal Investigator — Intermountain Medical Center; Stephen Archer, MD, Principal Investigator — University of Chicago; Andrew Kao, MD, Principal Investigator — Mid America Heart Institute, Saint Luke's Hospital; Paul J. Hauptman, MD, Principal Investigator — St. Louis University Hospital; Jill Kalman, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Douglas W. Losordo, MD, Principal Investigator — Northwestern University; Eric J. Eichhorn, MD, FACC, Principal Investigator — Cardiopulmonary Research Science and Technology Institutte, Medical City Dallas Hospital; Stephanie H. Dunlap, DO, Principal Investigator — University of Cincinnati; Vinay Thohan, MD, Principal Investigator — Wake Forest University; Maryl R. Johnson, MD, Principal Investigator — University of Wisconsin, Madison; Mark Dunlap, MD, Principal Investigator — MetroHealth Medical Center; Joaquin E. Cigarroa, MD, Principal Investigator — Oregon Health and Science University; Dinesh K. Gupta, MD, Principal Investigator — Tennessee Center for Clinical Trials, Harton Regional Medical Center; Marc Klapholz, MD, Principal Investigator — University of Medicine and Dentistry of New Jersey; Guillermo Torre, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (22):
- United States (22):
  - University of California at San Diego Medical Center, San Diego, California
  - San Diego Cardiac Center, San Diego, California
  - Shands Hospital at University of Florida, Gainesville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Mid America Heart Institute, Saint Luke's Hospital, Kansas City, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Columbia University Hospital, New York, New York
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Presbyterian-Shadyside Hospital, Pittsburgh, Pennsylvania
  - Tennessee Center for Clinical Trials & Harton Regional Medical Center, Tullahoma, Tennessee
  - Cardiopulmonary Research Science and Technology Institute, Medical City Dallas Hospital, Dallas, Texas
  - Methodist Hospital, Houston, Texas
  - Intermountain Medical Center, Murray, Utah
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Horowitz JD, Rosenson RS, McMurray JJ, Marx N, Remme WJ. Clinical Trials Update AHA Congress 2010. Cardiovasc Drugs Ther. 2011 Feb;25(1):69-76. doi: 10.1007/s10557-011-6285-9. PMID 21340529
- [Background] Hajjar RJ, Zsebo K, Deckelbaum L, Thompson C, Rudy J, Yaroshinsky A, Ly H, Kawase Y, Wagner K, Borow K, Jaski B, London B, Greenberg B, Pauly DF, Patten R, Starling R, Mancini D, Jessup M. Design of a phase 1/2 trial of intracoronary administration of AAV1/SERCA2a in patients with heart failure. J Card Fail. 2008 Jun;14(5):355-67. doi: 10.1016/j.cardfail.2008.02.005. Epub 2008 May 27. PMID 18514926
- [Result] Jaski BE, Jessup ML, Mancini DM, Cappola TP, Pauly DF, Greenberg B, Borow K, Dittrich H, Zsebo KM, Hajjar RJ; Calcium Up-Regulation by Percutaneous Administration of Gene Therapy In Cardiac Disease (CUPID) Trial Investigators. Calcium upregulation by percutaneous administration of gene therapy in cardiac disease (CUPID Trial), a first-in-human phase 1/2 clinical trial. J Card Fail. 2009 Apr;15(3):171-81. doi: 10.1016/j.cardfail.2009.01.013. PMID 19327618
- [Result] Jessup M, Greenberg B, Mancini D, Cappola T, Pauly DF, Jaski B, Yaroshinsky A, Zsebo KM, Dittrich H, Hajjar RJ; Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID) Investigators. Calcium Upregulation by Percutaneous Administration of Gene Therapy in Cardiac Disease (CUPID): a phase 2 trial of intracoronary gene therapy of sarcoplasmic reticulum Ca2+-ATPase in patients with advanced heart failure. Circulation. 2011 Jul 19;124(3):304-13. doi: 10.1161/CIRCULATIONAHA.111.022889. Epub 2011 Jun 27. PMID 21709064
- [Result] Zsebo K, Yaroshinsky A, Rudy JJ, Wagner K, Greenberg B, Jessup M, Hajjar RJ. Long-term effects of AAV1/SERCA2a gene transfer in patients with severe heart failure: analysis of recurrent cardiovascular events and mortality. Circ Res. 2014 Jan 3;114(1):101-8. doi: 10.1161/CIRCRESAHA.113.302421. Epub 2013 Sep 24. PMID 24065463

RESULTS

PARTICIPANT FLOW:
Groups:
- MYDICAR® Very Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1.4E11 DNAase resistant particles (DRP) administered by antegrade epicardial coronary artery infusion.
  This arm was included only in the Phase I open-label dose-escalation period.
- MYDICAR® Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 6E11 DNAase resistant particles (DRP) administered by antegrade epicardial coronary artery infusion.
- MYDICAR® Mid Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 3E12 DNAase resistant particles (DRP) administered by antegrade epicardial coronary artery infusion.
- MYDICAR® High Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1E13 DNAase resistant particles (DRP) administered by antegrade epicardial coronary artery infusion.
- Placebo: Single dose of placebo administered by antegrade epicardial coronary artery infusion.
  The placebo arm was included only in the Phase 2 randomized double-blind period.
Period: Phase I: Open-label Dose-escalation
Arm/Group | MYDICAR® Very Low Dose | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Started | 3 | 3 | 3 | 3 | 0
Completed | 2 | 2 | 2 | 2 | 0
Not Completed | 1 | 1 | 1 | 1 | 0
Not completed — Received heart transplant | 1 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0
Not completed — Received left ventricular assist device | 0 | 0 | 1 | 1 | 0
Period: Phase 2: Randomized Double-blind
Arm/Group | MYDICAR® Very Low Dose | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Started | 0 | 8 | 8 | 9 | 14
Completed | 0 | 6 | 5 | 8 | 10
Not Completed | 0 | 2 | 3 | 1 | 4
Not completed — Received milrinone or dobutamine | 0 | 1 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 1
Not completed — Received a heart transplant | 0 | 0 | 2 | 0 | 1
Not completed — Received left ventricular assist device | 0 | 0 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline data are provided for subjects enrolled in the Phase 1 or Phase 2 trials.
Groups:
- Phase 1: MYDICAR® Very Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1.4E11 DRP administered by antegrade epicardial coronary artery infusion.
- Phase 1: MYDICAR® Low Dose; Phase 2: MYDICAR® Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 6E11 DRP administered by antegrade epicardial coronary artery infusion.
- Phase 1: MYDICAR® Mid Dose; Phase 2: MYDICAR® Mid Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 3E12 DRP administered by antegrade epicardial coronary artery infusion.
- Phase 1: MYDICAR® High Dose; Phase 2: MYDICAR® High Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1E13 DRP administered by antegrade epicardial coronary artery infusion.
- Phase 2: Placebo: Single dose of placebo administered by antegrade epicardial coronary artery infusion.
- Total: Total of all reporting groups
Arm/Group | Phase 1: MYDICAR® Very Low Dose | Phase 1: MYDICAR® Low Dose | Phase 1: MYDICAR® Mid Dose | Phase 1: MYDICAR® High Dose | Phase 2: MYDICAR® Low Dose | Phase 2: MYDICAR® Mid Dose | Phase 2: MYDICAR® High Dose | Phase 2: Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 8 | 8 | 9 | 14 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (7.02) | 55.7 (4.51) | 48.0 (8.54) | 58.77 (19.01) | 60.3 (10.27) | 63.9 (8.85) | 56.6 (13.96) | 61.0 (11.94) | 60.5 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 1 | 1 | 0 | 3 | 1 | 8
  Male | 3 | 2 | 2 | 2 | 7 | 8 | 6 | 13 | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 6
  White | 3 | 3 | 1 | 3 | 8 | 8 | 6 | 13 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Incidence of Treatment-emergent Adverse Events (TEAE) at 12 Months
Description: Includes all adverse events that occurred from the time of first infusion of the investigational product or placebo to the 12-month visit. The category of "TEAEs related to the investigational product (IP)" includes TEAEs considered by the investigator to be possibly, probably, or definitely related to the IP.
Time Frame: 12 months
Population: This analysis was performed on the intention to treat population of the Phase 2 period, which included all patients randomized to treatment in the Phase 2 trial.
Measure: Number; unit: percentage of participants
Groups:
- MYDICAR® Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 6E11 DRP administered by antegrade epicardial coronary artery infusion.
- MYDICAR® Mid Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 3E12 DRP administered by antegrade epicardial coronary artery infusion.
- MYDICAR® High Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1E13 DRP administered by antegrade epicardial coronary artery infusion.
- Placebo: Single dose of placebo administered by antegrade epicardial coronary artery infusion.
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
percentage of participants
  Any TEAE | 100 | 100 | 88.9 | 92.9
  TEAEs related to the investigational product (IP) | 50 | 12.5 | 11.1 | 57.1
  TEAEs related to administration of the IP | 12.5 | 25 | 11.1 | 57.1
  Serious TEAEs | 62.5 | 50 | 33.3 | 64.3
  Serious TEAEs related to the IP | 0 | 0 | 0 | 21.4
  Serious TEAEs related to IP administration | 0 | 0 | 0 | 28.6

2. Primary Outcome: Phase 2: Length of Cardiovascular-related Hospitalizations at 6 Months
Description: Mean number of days in the hospital for cardiovascular-related complications. All hospitalizations were evaluated and classified by the blinded Clinical Endpoints Committee.
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
days | 0.3 (0.46) | 1.3 (2.55) | 0.2 (0.67) | 2.1 (2.92)
Statistical Analysis 1: Comparison: MYDICAR® High Dose vs Placebo; Test type: Superiority or Other; p = 0.078, t-test, 2 sided — The a priori threshold for statistical significance was P < 0.2. There were no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: MYDICAR® Mid Dose vs Placebo; Test type: Superiority or Other; p = 0.515, t-test, 2 sided — The a priori threshold for statistical significance was P < 0.2. There were no adjustments for multiple comparisons
Statistical Analysis 3: Comparison: MYDICAR® Low Dose vs Placebo; Test type: Superiority or Other; p = 0.098, t-test, 2 sided — The a priori threshold for statistical significance was P < 0.2. There were no adjustments for multiple comparisons

3. Primary Outcome: Phase 2: Change in Symptomatic Efficacy Domains From Baseline to Month 6: New York Heart Association (NYHA) Class and Minnesota Living With Heart Failure Questionnaire (MLWHFQ) Score
Description: NYHA classification is a symptomatic assessment in which the investigator evaluates subjects on a scale ranging from Class I (subjects with no limitation of activities, no symptoms from ordinary activities) to Class IV (subjects who should be at complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest).
  The MLWHFQ is a patient-reported quality of life (QoL) measure in which patients assess the impact of their heart condition on activities in the past month using a Likert scale ranging from 0 (no effect) to 5 (very much effect). Higher scores thus indicate a lower QoL. The maximum (worst) score is 105 and the minimum (best) score is 0.
  For both measures, changes from baseline with positive values indicate a worsening in symptoms and changes from baseline with negative values indicate an improvement in symptoms.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
units on a scale
  Change in NHYA class | -0.8 (0.71) | -0.8 (0.89) | -0.6 (0.73) | -0.2 (0.70)
  Change in MLWHFQ score | -7.6 (20.99) | 7.9 (27.28) | -10.3 (12.21) | 3.4 (36.00)

4. Primary Outcome: Phase 2: Change in 6-minute Walk Test (6MWT) From Baseline to Month 6
Description: The 6MWT measures the distance walked in meters during a 6-minute test. Higher values indicate a better functional status. Changes from baseline with negative values indicate a worsening in function and changes from baseline with positive values indicate an improvement in function.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
meters | 13.0 (61.40) | -59.5 (213.64) | 1.0 (99.69) | -86.6 (164.30)

5. Primary Outcome: Phase 2: Change in Peak Maximum Oxygen Consumption (VO2) From Baseline to Month 6
Description: Peak VO2 is a measure of maximal oxygen consumption during cardiopulmonary exercise testing; this study used the modified Naughton treadmill protocol. Higher values indicate a better functional status. Changes from baseline with negative values indicate a worsening in function and changes from baseline with positive values indicate an improvement in function.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/kg per minute
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
mL/kg per minute | -0.73 (4.88) | -1.07 (5.076) | -0.43 (0,802) | -2.10 (4.462)

6. Primary Outcome: Phase 2: Change in Absolute Levels of N-terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) From Baseline to Month 6
Description: NT-proBNP is a biomarker for heart failure. Increased levels of this biomarker are associated with increased mortality and cardiovascular hospitalization in patients with heart failure.
Time Frame: Baseline to 6 months
Population: This analysis was performed on the intention to treat population of the Phase 2 period, which included all patients randomized to treatment in the Phase 2 trial. NT-proBNP data were not available for 1 patient in the MYDICAR high dose group.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 14
pg/mL | 694.1 (1444.94) | 2073.1 (4224.22) | -13.5 (928.48) | 5540.0 (11,873.46)

7. Other Pre Specified Outcome: Phase 2: Length of Cardiovascular-related Hospitalizations at 12 Months
Description: as for outcome 2
Time Frame: 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
days | 10.1 (12.71) | 7.4 (11.80) | 0.4 (1.33) | 4.5 (5.80)

8. Other Pre Specified Outcome: Phase 2: Change in Symptomatic Efficacy Domains From Baseline to Month 12: New York Heart Association (NYHA) Class and Minnesota Living With Heart Failure Questionnaire (MLWHFQ) Score
Description: as for outcome 3
Time Frame: Baseline to 12 months
Population: This analysis was performed on the intention to treat population, which included all patients randomized to treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
units on a scale
  Change in NHYA class | -0.1 (0.99) | 0.1 (0.83) | -0.3 (0.71) | 0.1 (0.73)
  Change in MLWHFQ score | 24.4 (37.3) | 22.5 (32.56) | 0.1 (23.80) | 14.7 (34.89)

9. Other Pre Specified Outcome: Phase 2: Change in 6-minute Walk Test (6MWT) From Baseline to Month 12
Description: as for outcome 4
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
meters | -167.9 (191.02) | -115.9 (226.56) | -23.7 (151.08) | -120.4 (181.41)

10. Other Pre Specified Outcome: Phase 2: Change in Peak Maximum Oxygen Consumption (VO2) From Baseline to Month 12
Description: as for outcome 5
Time Frame: Baseline to 12 months
Population: This analysis was performed on the intention to treat population of the Phase 2 period, which included all patients randomized to treatment in the Phase 2 trial. Peak VO2 data were not available for one patient in the placebo group.
Measure: Mean (Standard Deviation); unit: mL/kg per minute
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 13
mL/kg per minute | -5.00 (4.733) | -3.31 (5.473) | -1.57 (3.677) | -2.75 (5.084)

11. Other Pre Specified Outcome: Phase 2: Change in Absolute Levels of N-terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) From Baseline to Month 12
Description: as for outcome 6
Time Frame: Baseline to 12 months
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 8 | 14
pg/mL | 3689.1 (5109.27) | 8440.4 (11270.44) | 1756.3 (4331.00) | 11464.3 (16866.55)

12. Post Hoc Outcome: Phase 2: Selected Clinical Outcomes During 12-month Study Period
Description: Incidences of key clinical endpoints as adjudicated by the blinded Clinical Endpoint Committee.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
percentage of participants
  Fatal cardiovascular event | 12.5 | 0 | 0 | 7.1
  Worsening heart failure | 50.0 | 37.5 | 22.2 | 50.0
  Myocardial infarction | 0 | 0 | 0 | 14.3
  Heart failure-related hospitalization | 50.0 | 37.5 | 22.2 | 42.9
  Silent myocardial infarction | 0 | 0 | 0 | 0
  Receipt of left ventricular assist device | 0 | 12.5 | 0 | 14.3
  Heart transplant | 0 | 25.0 | 11.1 | 7.1

13. Other Pre Specified Outcome: Phase 2: Change in Percentage of Blood Ejected From the Left Ventricle (LV) (i.e., Left Ventricular Ejection Fraction [LVEF]) From Baseline to Month 12
Description: Contrast echocardiography was used to determine LVEF. Increases in LVEF are associated with reduced mortality. Changes from baseline with positive values indicate an improvement in heart function and changes from baseline with negative values indicate a worsening of heart function.
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of blood ejected from the LV
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
Percentage of blood ejected from the LV | -6.5 (7.26) | -5.6 (10.52) | 0.3 (8.87) | -2.5 (9.96)

14. Primary Outcome: Phase 2: Change in Percentage of Blood Ejected From the Left Ventricle (LV) (i.e., Left Ventricular Ejection Fraction [LVEF]) From Baseline to Month 6
Description: as for outcome 13
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of blood ejected from the LV
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
Percentage of blood ejected from the LV | 0.0 (1.87) | -1.5 (6.35) | -0.7 (3.76) | -2.1 (6.90)

15. Primary Outcome: Phase 2: Change in Absolute Left Ventricular End Systolic Volume (LVESV) Frm Baseline to Month 6
Description: Contrast echocardiography was used to determine LVESV. Decreases in LVESV are associated with reduced mortality. Changes from baseline with positive values indicate a worsening in heart function and changes from baseline with negative values indicate an improvement in symptoms.
Time Frame: Baseline to 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
mL | 0.4 (26.16) | 10.5 (45.91) | -9.6 (27.55) | 18.2 (39.45)

16. Other Pre Specified Outcome: Phase 2: Change in Absolute Left Ventricular End Systolic Volume (LVESV) From Baseline to Month 12
Description: as for outcome 15
Time Frame: Baseline to 12 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Number analyzed (Participants) | 8 | 8 | 9 | 14
mL | 40.7 (59.79) | 66.8 (103.12) | 9.9 (49.27) | 37.7 (69.09)

17. Other Pre Specified Outcome: Phase 1 and Phase 2: All Subject Deaths Through 36 Months
Description: All subject deaths that occurred during the 12-month study or the 24-month follow-up in subjects enrolled in either the Phase 1 or Phase 2 trial. Events occurring after early termination from the trial are listed as occurring during long-term follow-up, but may have been within 12 months. Specifically, two cardiovascular (CV) deaths in placebo subjects occurred following early study termination, but within 12 months of study initiation. These deaths are therefore included under "Deaths within 12 months" but also listed as "Cardiovascular deaths in long-term follow-up." Accordingly, the number of "Cardiovascular deaths in long-term follow-up" for the placebo group is greater than the number of "Deaths after 12 months," as 2 of the deaths occurred within 12 months but after early termination.
Time Frame: 36 months
Population: Includes all participants enrolled in the Phase 1 or Phase 2 trial. Events occurring after early termination are listed under long-term follow-up. The number of "CV deaths in long-term follow-up" for the placebo group is greater than the number of "Deaths after 12 months," as 2 deaths occurred within 12 months but after early termination.
Measure: Number; unit: participants
Groups:
- MYDICAR® Very Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1.4E11 DRP administered by antegrade epicardial coronary artery infusion.
- All MYDICAR®: All participants who received a single infusion of MYDICAR® at any dose during the Phase 1 or Phase 2 studies.
Arm/Group | MYDICAR® Very Low Dose | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | All MYDICAR® | Placebo
Number analyzed (Participants) | 3 | 11 | 11 | 12 | 37 | 14
participants
  Deaths within 12 months | 0 | 2 | 0 | 0 | 2 | 3
  Deaths after 12 months | 1 | 2 | 3 | 2 | 8 | 3
  Cardiovascular deaths on study | 0 | 2 | 0 | 0 | 2 | 1
  Cardiovascular deaths in long-term follow-up | 1 | 2 | 1 | 2 | 6 | 4
  All deaths during 36 months | 1 | 4 | 3 | 2 | 10 | 6

ADVERSE EVENTS:
Time Frame: All treatment-emergent adverse events (TEAEs) that occurred from the time of first infusion of the investigational product or placebo through the 12-month visit.
Description: These data include all TEAEs occurring during the Phase 1 or Phase 2 parts of this study.
Groups:
- MYDICAR® Very Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 1.4E11DRP administered by antegrade epicardial coronary artery infusion.
- MYDICAR® Low Dose: Single dose of MYDICAR®, a viral vector (adeno-associated virus serotype 1 [AAV1]) carrying the gene for sarcoplasmic reticulum Ca++-adenosine triphosphatase (SERCA2a), at a dose of 6E11DRP administered by antegrade epicardial coronary artery infusion.
Arm/Group | MYDICAR® Very Low Dose | MYDICAR® Low Dose | MYDICAR® Mid Dose | MYDICAR® High Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 2/3 | 6/11 | 5/11 | 4/12 | 9/14
Other Adverse Events (participants affected / at risk) | 2/3 | 11/11 | 11/11 | 11/12 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MYDICAR® Very Low Dose (N=3) | MYDICAR® Low Dose (N=11) | MYDICAR® Mid Dose (N=11) | MYDICAR® High Dose (N=12) | Placebo (N=14)
Cardiac failure (Cardiac disorders) | 0 | 1 | 4 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 1 | 1 | 3
Cardiac failure acute (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiorenal syndrome (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Brain stem stroke (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Catheterization cardiac (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0
Heart transplant (Surgical and medical procedures) | 1 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Colonoscopy (Investigations) | 0 | 0 | 0 | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sudden death (General disorders) | 0 | 1 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MYDICAR® Very Low Dose (N=3) | MYDICAR® Low Dose (N=11) | MYDICAR® Mid Dose (N=11) | MYDICAR® High Dose (N=12) | Placebo (N=14)
Anemia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 2 | 2 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 3 | 0 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 3 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 2 | 2 | 2 | 2
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0
External ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Catheter site hematoma (General disorders) | 0 | 0 | 1 | 0 | 0
Catheter site hemorrhage (General disorders) | 0 | 0 | 1 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 1
Chest pain (General disorders) | 0 | 1 | 0 | 3 | 1
Chills (General disorders) | 0 | 1 | 1 | 0 | 1
Fatigue (General disorders) | 1 | 3 | 2 | 2 | 4
Feeling jittery (General disorders) | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 1
Edema (General disorders) | 0 | 0 | 1 | 0 | 0
Edema peripheral (General disorders) | 0 | 1 | 0 | 1 | 0
Puncture site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 2
Venipuncture site thrombosis (General disorders) | 0 | 1 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 2 | 0 | 1 | 2
Candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Central line infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Gastric ulcer Helicobacter (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 0 | 3 | 1 | 1 | 2
Viral infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2
Eye injury (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 1 | 1 | 0 | 0
Blood creatinine phosphokinase MB increased (Investigations) | 0 | 2 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 1
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0
Carcinoembryonic antigen increased (Investigations) | 0 | 0 | 0 | 0 | 1
Gallop rhythm present (Investigations) | 0 | 0 | 0 | 0 | 2
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1 | 1
International normalized ratio increased (Investigations) | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1 | 0 | 1 | 1
Mean cell volume increased (Investigations) | 0 | 0 | 0 | 1 | 0
Muscle enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 0 | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Weight increased (Investigations) | 0 | 1 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 2 | 1 | 2 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypervolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 2 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0
Hypovolemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1
Asterixis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 1 | 4
Dizziness postural (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypoesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Neurological symptom (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Nystagmus (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Restless leg syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 2
Bruxism (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 3
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Somnambulism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Azotemia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2
Hematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1
Breast disorder (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Gynecomastia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0
Variocele (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 1
Dyspnea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 1
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Orthopnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 0
Sleep apnea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Hemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Rash generalized (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Cataract operation (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 1 | 2 | 1

LIMITATIONS AND CAVEATS:
Limitations of this study include its small sample size and the inability to conclusively prove that the delivered gene was responsible for the observed clinical effects. Larger confirmatory trials are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days